CLINICAL TRIAL: NCT03638401
Title: Epidural vs. Wound Catheter Following Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Other
Other Study IDs: RL14/11048
Record Dates: First submitted 2015-05-18; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Transplant Surgery

ARMS (2):
- Standard treatment (No Intervention)
- Intervention arm (Active Comparator)
  Interventions: Procedure: This arm will received perioperative transversus abdominis plane (TAP) block followed by continuous infusion of local anaestheic by wound catheters and an IV morphine PCA.

INTERVENTIONS:
Procedure: This arm will received perioperative transversus abdominis plane (TAP) block followed by continuous infusion of local anaestheic by wound catheters and an IV morphine PCA. — This arm will received perioperative transversus abdominis plane (TAP) block followed by continuous infusion of local anaestheic by wound catheters and an IV morphine PCA.
  Arms: Intervention arm

SUMMARY:
Good postoperative pain control after any major surgery allows early mobilization, minimises postoperative complications and reduces patient distress. Multiple different methods of delivering analgesia have been described.

This study aims to compare postoperative pain control between patients with epidural analgesia versus the combination of continuous infiltration of local anaesthetic with wound catheters, TAP block and IV PCA with opiate analgesia following open liver resection. The investigators expect that pain control will be similar between the two groups but that the utilization of wound catheters will confer benefit due to the lack of systemic side effects associated with epidural analgesia

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled to undergo an open liver resection at this hospital will be eligible to participate.

Exclusion Criteria:

* Patients with a contraindication to either epidural or wound catheter
* Inability to give written, informed consent
* Aged less than 18 years old
* Liver resection combined with a secondary surgical procedure
* Body mass index of <18 or >40
* Pregnancy or lactation
* A history of chronic pain requiring regular opioid analgesia
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-05 (Actual)

PRIMARY OUTCOMES:
The length of hospital stay following open liver resection | 6 months (or length of the study)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom